CLINICAL TRIAL: NCT04524585
Title: Partial Neuromuscular Blockade in Acute Hypoxemic Respiratory Failure
Acronym: PNEUMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-5975
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Insufficiency; Neuromuscular Blockade; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — cisatracurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partial NMB (Experimental)
  Interventions: Drug: Cisatracurium

INTERVENTIONS:
Drug: Cisatracurium — Cisatracurium will be infused to achieve Pocc targets after ensuring adequate sedation. Sedation will be titrated to avoid dyspnea, assessed with P0.1 targets between -1.5 and -3.5 cmH2O and Mechanical Ventilation Respiratory-Distress Observation Scale (MV-RDOS) ≤ 3. If there is no sign of dyspnea or discomfort based on P0.1, MV-RDOS, hemodynamics and the train-of-four ratio is ≥ 60% (compatible with ability to interact using peripheral muscles), sedation will be carefully reduced. After establishing a sedation and NMB strategy at which safe spontaneous breathing is achieved, we will seek to determine whether these targets can be maintained over a 48-hour period or until hypoxemia is resolved (FiO2 ≤ 40% on PEEP ≤ 8 cmH2O), whichever occurs first.

SUMMARY:
PNEUMA is a preliminary safety and feasibility trial of a novel approach to the titration of neuromuscular blockade (NMB) to safe spontaneous breathing in patients with moderate to severe acute hypoxemic respiratory failure (AHRF) supported with invasive mechanical ventilation.

DETAILED DESCRIPTION:
Controlling respiratory effort in patients with AHRF can be challenging, as they often exhibit a very high respiratory drive despite receiving high doses of sedatives. Consequently, these patients usually receive full neuromuscular blockade, with the goal to avoid such injurious respiratory efforts. Unfortunately, full neuromuscular blockade is not without complications. To address this issue, the use of partial neuromuscular blockade has been proposed as a strategy to maintain respiratory muscle activity while providing lung protective ventilation.

The objective of this study is to demonstrate the safety and feasibility of safe spontaneous breathing using partial NMB in moderato to severe AHRF patients supported with invasive mechanical ventilation.

Once adequate sedation has been ensured, an infusion of cisatracurium will be started to maintain spontaneous breathing with moderate levels of inspiratory effort, defined by expiratory occlusion pressure (Pocc) between -5 and -15 cmH2O. After establishing a sedation and NMB dosing regimen at which safe spontaneous breathing is achieved, we will document whether these targets can be maintained over a 48-hour period.

On December 11 2025, this study has been amended to broaden eligibility criteria from patients with acute respiratory distress syndrome supported on extracorporeal membrane oxygenation (ECMO) to patients with AHRF supported with invasive mechanical ventilation or with venovenous-ECMO. Additionally, the study intervention duration was extended from 24 hours to 48 hours or until hypoxemia is resolved (FiO2 ≤ 40% on PEEP ≤ 8 cmH2O), whichever occurs first. Finally, the study intervention was modified to remove the use of esophageal balloon, and to include sedation and neuromuscular blockade titration targeting Pocc between -5 to -15 cmH2O and according to predefined safety criteria assessed using train of four, respiratory drive and comfort assessments. A total of 15 patients will be enrolled after the amendment, in addition to the 8 patients already enrolled, for a total of 23 patients. Going forward, only patients in whom the intervention is initiated will count toward the study sample size.

ELIGIBILITY:
Inclusion Criteria:

Patients supported on invasive mechanical ventilation for moderate to severe AHRF (PaO2/FiO2 < 150 mm Hg or FiO2 ≥ 60% with an SpO2 ≤ 97% or receiving venovenous extracorporeal membrane oxygenation)

Exclusion Criteria:

1. Contraindication to neuromuscular blockade (allergy, history of malignant hyperthermia)
2. Contraindication to ulnar nerve stimulation (bilateral peripheral neuropathy, skin burns on both wrists)
3. Previous history of a formally diagnosed neuromuscular disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients achieving and maintaining targeted expiratory occlusion pressure (Pocc) | Assessed for 48 hours after study intervention initiation

SECONDARY OUTCOMES:
Rates of serious adverse events | Assessed for 48 hours after study intervention initiation
Paralysis Recall | Assessed after 48 hours of the study intervention, as soon as the patient is extubated and oriented.
  Evaluted using the modified Brice questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada